CLINICAL TRIAL: NCT01325233
Title: The Pilot Clinical Study of PG2 Injection on Hemorrhagic Stroke
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP018
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Hemorrhagic Stroke
Keywords: Astragulus polysaccharides; Hemorrhagic stroke
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PG2 Injection (Experimental): Powder for Injection, 500 mg PG2/500 ml normal saline, tiw, 2 weeks
  Interventions: Drug: PG2
- Placebo (Placebo Comparator): Powder for Injection, 500 ml normal saline, tiw, 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PG2 — Powder for Injection, 500 mg PG2/500 ml normal saline, tiw, 2 weeks
  Arms: PG2 Injection
Drug: Placebo — 500 ml normal saline, tiw, 2 weeks
  Arms: Placebo

SUMMARY:
Astragalus membranaceus (AM) is used to treat stroke for a long time, and a number of studies have shown that AM can reduce cerebral infarction area and has anti-oxidation activity. PG2, a sterile powder of polysaccharides isolated from the root of astragulus (Huang-Chi) for intravenous injection, has been approved as a botanical drug by TFDA. Hemorrhagic stroke will induce secondary peri-blood clot edema and that may increase intracranial pressure to exacerbate clinical symptom. Therefore, the purpose of the present study was to investigate the efficacy of PG2 on hemorrhagic stroke.

DETAILED DESCRIPTION:
This will be a double-blind, randomized, placebo-controlled study. An estimated 60 (at least 48 evaluable) first hemorrhagic stroke patients will be randomly divided into the control and treatment groups. Each group will be treated as follows: 1) control group will accept placebo t.i.w treatment for 14 days from second day of admission, in addition to standard ordinary treatment.; 2) treatment group will accept PG2 t.i.w treatment for 14 days from second day of admission, in addition to standard ordinary treatment. Inflammatory index including the levels of C-Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), S-100 protein, IL-1, IL-6, and TNF-beta levels will be measured and clinical symptoms including Glasgow outcome scale (GOS), modified rankin scale (MRS), Functional Independence Measure (FIM) and Barthel Index (BI) will be evaluated during this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who confirmed diagnosis of first spontaneous hemorrhagic stroke
* Patients with hemorrhagic stroke in Putamen
* Patients who admitted to the hospital within 24 hours of onset of hemorrhagic stroke
* Patients who signed the informed consent form

Exclusion Criteria:

* Patient with hemorrhage in the area out of Putamen or primary subarachnoid hemorrhage, Arteriovenous malformation (AVM) or brain tumor hemorrhage
* Patient who performed craniotomy
* Patient who suffering from cirrhosis, uremia with dialysis, bleeding tendency, severe cardiopulmonary disease or mental disorders would be unable to comply with the study by investigators' decision.
* Patients have enrolled or have not yet completed other investigational drug trials within 1 month before screening.
* Female patients are pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | FIM will be evaluated on day 1 (baseline, before study drug treatment), day 7, day 28 and day 84.

SECONDARY OUTCOMES:
Other clinical symptoms including Glasgow outcome scale (GOS), modified rankin scale (MRS), and Barthel Index (BI) | These clinical symptoms will be evaluated on on day 1 (baseline, before study drug treatment), day 7, day 28 and day 84.
Inflammatory index including C-Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), S-100 protein, IL-1, IL-6, and TNF-beta levels. | These index will be detected on day 1 (baseline, before study drug treatment), day 4 and day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Chung CC Chen, MD, Principal Investigator — China Medical University Hospital, Taichung, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan